CLINICAL TRIAL: NCT02310087
Title: Effect of Oral Administration of Astaxanthin on Semen Quality, Fertilization and Embryo Development in Assisted Reproduction Techniques Procedures
Brief Title: Oral Astaxanthin and Semen Quality, Fertilization and Embryo Development in Assisted Reproduction Techniques Procedures
Acronym: Astax-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Bojana Pinter, Assoc. Prof., MD, PhD, Spec in Ob/Gyn, MS (Econ), University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMCLjubljana-20140041
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Infertility, Male
Keywords: male infertility; spermatogenesis; antioxidants; DNA damage; mitochondrial membrane potential; apoptosis
MeSH Terms: conditions — Infertility, Male | interventions — astaxanthine; Vitamin E

STUDY DESIGN:
Intervention Model Description: Eighty infertile men with OAT were randomly assigned to receive either daily 16 mg of astaxanthin and 40 mg of vitamin E in capsules or placebo. At baseline and after three months of treatment semen quality was assessed according to the WHO guidelines. The sperm concentration, motility and morphology were determined by standard microscopic analyses. Sperm DNA fragmentation was evaluated using a TUNEL assay . Mitochondrial membrane potential was measured by means of 3,3'-dihexyloxacarbocyanine iodide (DiOC6) staining as an indicator of mitochondrial membrane integrity and the mitochondrial potential capacity to generate ATP by oxidative phosphorylation. The serum level of FSH was measured by a solid-phase, two-site chemiluminescent immunometric assay.
Who Masked: Participant, Care Provider, Investigator
Masking Description: no other masking
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- astaxanthin with vitamin E (Active Comparator): The participants in the study group will be given perorally four tablets of 4 mg astaxanthin with 10 mg vitamin E (Astasan, Sensilab, Slovenia) daily, taken in single daily dose. The total daily dose will be 16 mg astaxanthin with 40 mg vitamin E. The product will be taken for three months continuously.
  Interventions: Dietary Supplement: astaxanthin with vitamin E
- placebo (Placebo Comparator): The participants in the control group will be given perorally four tablets of placebo daily taken in single daily dose. The placebo tablets are of the same size and colour as the study tablets and were produced by manufacturer of Astasan, Sensilab, Slovenia. The placebo will be taken for three months continuously.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: astaxanthin with vitamin E — Four tablets of 4 mg astaxanthin with 10 mg vitamin E daily, taken at once. Daily dose is 16 mg astaxanthin with 40 mg vitamin E. Continuously for three months.
  Other Names: Astasan, Sensilab, Slovenia
  Arms: astaxanthin with vitamin E
Other: Placebo — Four tablets of placebo daily, taken at once. Continuously for three months.
  Arms: placebo

SUMMARY:
The purpose of the study is to determine whether administration of dietary supplement of astaxanthin with vitamin E improves the quality of sperm, fertilization and embryo development in Assisted Reproduction Techniques (ART) procedures.

DETAILED DESCRIPTION:
In the study male patients diagnosed with oligoasthenozoospermia - with an abnormal sperm concentration and motility, irrespective of the morphology of spermatozoa - treated with their female partner with assisted reproduction techniques (ISCI) will be included. In the double blind study male patients will be given astaxanthin with vitamin E (study group, 40 patients) or placebo (control group, 40 patients) for three months prior to ART. In the study and the control group the quality of sperm (spermiogram), DNA fragmentation and mitochondrial membrane potential of semen before and after the dietary supplementation will be evaluated. In the ART procedure (ICSI) the fertilization rate, the quality of embryos, pregnancy rates and miscarriages rates in 1st trimester will be compared between the study and control group.

ELIGIBILITY:
Inclusion Criteria:

* oligoasthenozoospermia with of without teratozoospermia by WHO criteria from the year 2010
* fresh semen
* female partner younger than 38 years
* idiopathic or tubal infertility in female partners
* at least 4 oocytes retrieved in previous ovarian punction in ART cycle, if previously performed
* 1st, 2nd or 3rd cycle of ART

Exclusion Criteria:

* genetic indication for ART procedure
* donated semen
* polycystic ovary syndrome in female partner
* dietary supplementation intake of antioxidants (selenium, zink, vitamin E, vitamin C, vitamin A) in male participant in the last three months
* smoking in male participant >20 cigarettes per day

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
semen quality | three months
  In semen quality the spermiogram, DNA fragmentation and mitochondrial membrane potential before and after the intervention will be evaluated. The DNA fragmentation will be evaluated by terminal deoxynucleotidyl transferase-mediated deoxyuridine triphosphate (dUTP)-biotin nick end labeling (TUNEL) method, and mitochondrial membrane potential with carbocyanine fluorochrome DiOC6.

SECONDARY OUTCOMES:
follicle stimulating hormone (FSH) | three months
  FSH levels in before and after the intervention will be evaluated in infertile men with oligoasthenozoospermia.
fertilization and embryo development in Assisted Reproduction Techniques (ART) | six months
  Fertilization rates and the quality of embryo development on day 3 in ICSI procedure in infertile couples will be determined after the three months of dietary supplementation of astaxanthin with vitamin E taken by infertile men with oligoasthenozoospermia.
pregnancy rates and miscarriage rates in 1st trimester after ART | nine months
  Pregnancy rates and miscarriage rates in 1st trimester after ART will be determined after the three months of dietary supplementation of astaxanthin with vitamin E taken by infertile men with oligoasthenozoospermia.

CONTACTS AND LOCATIONS:
Overall Officials: Bojana Pinter, MD, PhD, Principal Investigator — Division of Ob/Gyn, University Medical Centre Ljubljana, Slovenia
Locations (1):
- Division of Ob/Gyn, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analysed during the current study could not be publicly available because they are in the Slovene language. Unauthorised translation may lead to data misunderstanding or misinterpretation.

REFERENCES:
- [Background] Imamovic Kumalic S, Pinter B. Review of clinical trials on effects of oral antioxidants on basic semen and other parameters in idiopathic oligoasthenoteratozoospermia. Biomed Res Int. 2014;2014:426951. doi: 10.1155/2014/426951. Epub 2014 Mar 31. PMID 24800224
- [Background] Yuan JP, Peng J, Yin K, Wang JH. Potential health-promoting effects of astaxanthin: a high-value carotenoid mostly from microalgae. Mol Nutr Food Res. 2011 Jan;55(1):150-65. doi: 10.1002/mnfr.201000414. Epub 2010 Nov 18. PMID 21207519
- [Background] Agarwal A, Nallella KP, Allamaneni SS, Said TM. Role of antioxidants in treatment of male infertility: an overview of the literature. Reprod Biomed Online. 2004 Jun;8(6):616-27. doi: 10.1016/s1472-6483(10)61641-0. PMID 15169573
- [Background] Higuera-Ciapara I, Felix-Valenzuela L, Goycoolea FM. Astaxanthin: a review of its chemistry and applications. Crit Rev Food Sci Nutr. 2006;46(2):185-96. doi: 10.1080/10408690590957188. PMID 16431409
- [Background] Comhaire FH, El Garem Y, Mahmoud A, Eertmans F, Schoonjans F. Combined conventional/antioxidant "Astaxanthin" treatment for male infertility: a double blind, randomized trial. Asian J Androl. 2005 Sep;7(3):257-62. doi: 10.1111/j.1745-7262.2005.00047.x. PMID 16110353
- [Background] Franco JG Jr, Baruffi RL, Mauri AL, Petersen CG, Oliveira JB, Vagnini L. Significance of large nuclear vacuoles in human spermatozoa: implications for ICSI. Reprod Biomed Online. 2008 Jul;17(1):42-5. doi: 10.1016/s1472-6483(10)60291-x. PMID 18616888
- [Background] Chemes EH, Rawe YV. Sperm pathology: a step beyond descriptive morphology. Origin, characterization and fertility potential of abnormal sperm phenotypes in infertile men. Hum Reprod Update. 2003 Sep-Oct;9(5):405-28. doi: 10.1093/humupd/dmg034. PMID 14640375
- [Background] Virro MR, Larson-Cook KL, Evenson DP. Sperm chromatin structure assay (SCSA) parameters are related to fertilization, blastocyst development, and ongoing pregnancy in in vitro fertilization and intracytoplasmic sperm injection cycles. Fertil Steril. 2004 May;81(5):1289-95. doi: 10.1016/j.fertnstert.2003.09.063. PMID 15136092
- [Background] Marchetti C, Obert G, Deffosez A, Formstecher P, Marchetti P. Study of mitochondrial membrane potential, reactive oxygen species, DNA fragmentation and cell viability by flow cytometry in human sperm. Hum Reprod. 2002 May;17(5):1257-65. doi: 10.1093/humrep/17.5.1257. PMID 11980749